CLINICAL TRIAL: NCT06935383
Title: Randomised EValuation of Therapies for microvAscuLar Injury in STEACS
Acronym: REVITALISE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CorFlow Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2503
Record Dates: First submitted 2025-04-17; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: STEMI (ST Elevation MI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Shame (Sham Comparator)
  Interventions: Device: Diagnostic sequence
- Treatment A (Experimental)
  Interventions: Device: Therapeutic sequence; Device: Diagnostic sequence
- Treatment B (Experimental)
  Interventions: Device: Therapeutic sequence; Device: Diagnostic sequence

INTERVENTIONS:
Device: Therapeutic sequence — the required dose of treatment is administered through the CoFI system
  Arms: Treatment A; Treatment B
Device: Diagnostic sequence — Diagnostic sequence to detect MVO

SUMMARY:
The goal of this interventional study is to evaluate if the CoFI system can act as a platform for intracoronary infusion of therapeutic agents to treat and relieve microvascular injury in ST Elevation Acute Coronary Syndrome (ACS) subjects diagnosed with MicroVascular Obstruction (MVO) after Primary Percutaneous Intervention (PPCI) and to quantify (identify) markers of treatment efficacy for CoFI mediated therapeutic agents infusion versus control.

The targeted population is subjects presenting with an ST elevation myocardial infarction and undergoing PPCI as per standard of care.

Enrolled STEMI subjects will be examined for MVO with the CoFI system. Primary endpoint of the study is EF by TTE at 6 months.

If detected with MVO with the CoFI system, the subjects will be randomized and will receive treatment with medicinal product(s).

ELIGIBILITY:
Inclusion Criteria:

CLINICAL criteria

1. Subjects age ≥18 years old
2. Ability to provide informed assent/consent to the study according to GCP, governing regulations and approved process
3. Infarct-related lesion in proximal or mid left anterior descending coronary artery
4. ECG evidence of acute anterior myocardial infarction with ST-elevation ≥ 2 mm (0.2 mV) in 2 or more contiguous anterior precordial ECG leads (one of which should be V2, V3, or V4) in men or ≥ 1.5 mm (0.15 mV) in women
5. Symptoms onset to balloon time consistent with myocardial ischemia (e.g. persistent chest pain, shortness of breath, nausea/vomiting, fatigue, palpitations or syncope) ≤ 6 h
6. Suitability for Primary PCI

   PPCI and Angiographic
7. Culprit lesion in the LAD that is suitable for stenting
8. COFI ballon can be placed according to IFU
9. Required stent diameter ≥ 2.75 mm and ≤ 5mm and stent length ≥ 15 mm

Exclusion Criteria:

CLINICAL criteria

1. Unconscious on presentation
2. Patients under judicial protection, legal guardianship or curatorship
3. Mental disorder or language barrier that precludes informed assent/consent GCP, governing regulations and approved process
4. Known severe kidney disease (estimated glomerular filtration rate (eGFR) < 30 ml/min) or on haemodialysis
5. Pericardial effusion (cardiac tamponade)
6. Cardiogenic shock and/or persistence of cardiogenic shock at completion of primary PCI. Cardiogenic shock defined as a. hypotension (systolic blood pressure below 100 mm Hg or an ongoing need for vasopressor support), and b. end-organ hypoperfusion with an arterial lactate level of 2.5 mmol/L or greater
7. Subject with previous MI and/or known cardiomyopathy (ischemic and non ischemic), ventricular pseudoaneurysm, ventricular Septal defect, severe mitral valve regurgitation (with or without papillary muscle rupture), severe known cardiac valvular stenosis or regurgitation, pericardial disease
8. Major bleeding ≤ 30d prior to intervention defined according to BARC 3-5
9. Major surgery ≤ 30d prior to intervention
10. History of stroke, TIA or reversible ischemic neurological deficit within last 6 months
11. Known coagulopathy
12. Treatment with oral anticoagulation therapy
13. Need for circulatory support or pre/intra-procedural ventilation
14. Patients with cardio-pulmonary resuscitated (CPR) cardiac arrest for more than 5 min
15. Heart failure with inotrope support and/or consideration for LVAD or heart transplant
16. Subject has other medical illness (e.g., cancer, dementia) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause non-compliance with the CIP, confound the data interpretation, or is associated with limited life expectancy of less than one year
17. Current participation in another clinical study
18. Known Pregnancy or breast feeding

    If CMRI substudy to be confirmed at the time of consent to the substudy:
19. Contraindication to CMRI

    1. Cardiac pacemaker or implantable defibrillator;
    2. Non-MRI compatible aneurysm clip;
    3. Neural Stimulator (i.e., TENS unit);
    4. Any implanted or magnetically activated device (insulin pump);
    5. Any type of non-MRI compatible ear implant;
    6. Metal shavings in the orbits;
    7. Any metallic foreign body, shrapnel, or bullet in a location which the physician feels would present a risk to the subject;
    8. Any history indicating contraindication to MRI
    9. Inability to follow breath hold instructions or to maintain a breath hold for >15 seconds; and
    10. Known hypersensitivity or contraindication to gadolinium contrast.

PPCI and Angiographic criteria 19. Functional coronary collateral supply (Rentrop grade 2/3) to the infarct-related artery 20. Unsuitable target vessel anatomy (excessive tortuosity, diffuse disease, or moderate/heavy calcification) preventing successful wiring with pressure wire 21. Cardiac condition preventing the use of the CoFI System 22. Any pre or post stenting condition that the physician believes requires a pharmacological iv or ic drug administration for a cardiac related condition to be administered before or during stenting, apart from standard of care administration of anaesthetics, heparin, nitrates or verapamil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Delta LVEF at post procedure and 6 months follow up visit | From enrollment to the 6 months follow up visit
  Absolute difference in left ventricular ejection fraction (LVEF) measured within 24 hours post-primary percutaneous coronary intervention (PPCI) and 6 months follow up, using transthoracic echocardiography (TTE) assessed blind to treatment group assignment.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Luigi De Maria, Principal Investigator — Oxford Heart Centre John Radcliffe Hospital Headley Way - OX3 9DU Oxford United Kingdom; Colin Berry, Principal Investigator — The Royal Golden Jubilee Hospital, Glasgow, Uk